CLINICAL TRIAL: NCT06510231
Title: Inspiratory Muscle Training in Heart Failure With Preserved Ejection Fraction
Brief Title: Inspiratory Muscle Training in HFpEF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Joshua R. Smith, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 24-003293; 1R01HL175086-01 (NIH)
Record Dates: First submitted 2024-07-15; First posted 2024-07-19 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inspiratory muscle training (IMT) group (Experimental): IMT performed at 40% maximal inspiratory pressure (MIP) for 30 minutes 7 days a week for 8 weeks.
  Interventions: Other: Inspiratory Muscle Training
- SHAM group (Sham Comparator): IMT performed at 2% maximal inspiratory pressure (MIP) for 30 minutes 7 days a week for 8 weeks.
  Interventions: Other: Inspiratory Muscle Training

INTERVENTIONS:
Other: Inspiratory Muscle Training — Inspiratory muscle training (IMT) targets the inspiratory muscles and is used to improve inspiratory muscle strength.

SUMMARY:
This study is being done to determine how inspiratory muscle training impacts inspiratory muscle function during exercise in heart failure patients.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 yrs of age
* Receiving SGLT2 inhibitors and spironolactone (and beta-blocker use for HFpEF patients with hypertension) for >3 months
* NYHA symptoms I-III
* Body mass index ≤40 kg/m2
* Currently non-smokers with <20 pack year history
* Able to exercise (i.e. without significant orthopedic limitations or musculoskeletal disorders limiting their ability to exercise)

Exclusion Criteria:

* Sustained ventricular tachycardia and/or ventricular fibrillation within 21 days of visit 1
* Second or third degree heart block
* Body mass index >40 kg/m2
* Current smokers and/or smoking history >20 pack years
* Pregnant women (testing will be done by research team if requested)
* Glomerular filtration rate of <30 mL/min/1.73m2 (initial screen via clinical record within the past 6 months and this will be assessed on Visit 1)
* Individuals who are not able to engage in exercise
* Uremia, history of allergy to iodides
* Peripheral artery disease
* Alanine transaminase and/or aspartate transaminase greater than 2 times the upper limit of normal (via clinical record within the past 6 months)
* Asthmatic patients with a low symptom perception and suffer frequency, severe exacerbations or with an abnormally low perception of dyspnea
* Ruptured eardrum or any other condition of the ear
* History of spontaneous pneumothorax or osteoporosis with a history of rib fractures
* History of lidocaine allergy.

For individuals agreeing to undergo dual energy x-ray absorptiometry (DEXA) scanning for measurement of body composition as part of their study visit, additional exclusion criteria apply: recently administered gastrointestinal contrast or radionuclides; severe degenerative changes or fracture deformity in measurement areas; or inability to attain correct position and/or remain motionless for the measurement period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2024-10-09 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Change in inspiratory muscle blood flow demand | Baseline, 8 weeks
  Inspiratory muscle blood flow demand will be measured via indocyanine green dye venous bolus injection. This will be measured in umol.

SECONDARY OUTCOMES:
Change in locomotor muscle blood flow | Baseline, 8 weeks
  Locomotor muscle blood flows will be measured via indocyanine green dye venous bolus injection. This will be measured in umol.
Change in exercise tolerance | Baseline, 8 weeks
  Exercise tolerance will be measured via submaximal exercise test. This will be measured in minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Smith, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No